CLINICAL TRIAL: NCT04165226
Title: Low Level Light Therapy and Fractional Carbon Dioxide Laser in the Treatment of Stria Alba: A Randomised Controlled Study
Brief Title: LLLT and Fractional CO2 Laser in the Treatment of Stria Alba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Marina Mikhail, Visiting resident, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMikhail
Record Dates: First submitted 2018-12-20; First posted 2019-11-15 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Striae; Albicantes
Keywords: Stria alba; Fractional CO2; Fractional carbon dioxide laser 00; Low level light therapy; Striae atrophicae; Infra red diode laser; 808 nm; 915 nm; 10600 nm
MeSH Terms: conditions — Striae Distensae | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low level light therapy (LLLT) (Active Comparator): Low level light therapy using 808/915 nm infra red diode laser
  Interventions: Device: Low level light therapy
- Fractional CO2 (Active Comparator): Fractional carbon dioxide laser 10600 nm
  Interventions: Device: Fractional CO2
- Combined fractional CO2 and LLLT (Active Comparator): Combined fractional CO2 laser and low level light therapy
  Interventions: Device: Combined fractional CO2 laser and low level light therapy

INTERVENTIONS:
Device: Low level light therapy — Patients will be offered 8 sessions of photobiomodulation using HPL Pagani Diode 808/915nm LLLT 3.2W (Fimad Elettromedicali SRL®, Catanzaro, Italy) with the parameters adjusted individually according to the surface area to be treated. Optimum dose is 10 joules/cubic centimeters. The patients will take 2 to3 sessions / week.
  Arms: Low level light therapy (LLLT)
Device: Fractional CO2 — Patients will be offered 2 sessions of fractional carbon dioxide laser on a 4 weeks interval. Topical anesthesia with pridocaine cream will be applied under occlusion for 30 - 60 minutes before the session.
  * Please update to the proper apparatus and parameters DEXA SmartXide DOT Fractional CO2 laser system 10600 nm (DEKA®, Florence, Italy) will be used with the following parameters adjusted individually to patients': power of 15-20 W, dwell time of 500-800 μs, spacing of 200-500 μm, and stack 2.
  Arms: Fractional CO2
Device: Combined fractional CO2 laser and low level light therapy — Combined treatment of both modalities (fractionational CO2 laser and low level light therapy). Please describe more....
  Arms: Combined fractional CO2 and LLLT

SUMMARY:
Stria alba (aka white or atrophic stretch marks) is a very common dermatologic condition that causes major psychological distress to those afflicted. We study the effect of low level light therapy using infra red diode 808/915 nm laser in comparison to fractional CO2 alone and combined both therapies.

DETAILED DESCRIPTION:
All patients will be subjected to the following:

* Written informed consent.
* Detailed history and clinical evaluation.

The treated areas will be photographed (in standardized settings of light and position) and measured in order to allow comparison and assessment of striae improvement following treatment.

Patients will be allocated according to randomization into one of 3 arms:

Arm A will be treated by fractional CO2 laser. Arm B will be treated by low level light therapy (LLLT). Arm C will be treated with a combination of fractional CO2 laser and LLLT.

Digital photographs will be taken for each patient, at the baseline and 1 and 3 months after last session and the width of the widest striae in each patient will be measured at the same time. Patients will be assessed before and after treatment by one unblinded and 2 blinded investigators to measure the clinical improvement on a 4-point scale by comparing the photographs. The criteria for evaluation using a quartile grading scale will be as follows; 0=no improvement, 1=mild improvement (<25%), 2=moderate improvement (26% - 50%), 3=good improvement (51% -75%), 4=excellent improvement (>76%).

In addition, a patient satisfaction score will be rated using the following scale; 0=not satisfied, 1=slightly satisfied, 2= satisfied, 3=very satisfied, 4=extremely satisfied as well as patients' satisfaction questionnaire (Yang and Lee; 2011).

ELIGIBILITY:
Inclusion Criteria:

* Subjects, above the age of 18 years old, with stria alba.
* Both genders.

Exclusion Criteria:

* Pregnant or lactating females.
* Subjects who were treated with any interventional procedure (lasers, radiofrequency, dermabrasion, microdermabrasion, or chemical peeling) within 6 months prior to the study.
* Subjects who applied topical corticosteroids, retinoid, vitamin C, or vitamin E within 3 months prior to the study.
* Subjects who orally took retinoids or corticosteroids within 3 months.
* Subjects who had a history of hypertrophic scar, keloid or immunosuppression or cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-24 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Comparative effectiveness of the 3 intervention groups as assessed by patient global assessment at month 3 (End of study) | 3 months
  Patients will be assessed before and after treatment by one unblinded and one blinded investigators to measure the clinical improvement on a 4-point scale by comparing the photographs. The criteria for evaluation using a quartile grading scale will be as follows; 0=no improvement, 1=mild improvement (<25%), 2=moderate improvement (26% - 50%), 3=good improvement (51% -75%), 4=excellent improvement (>76%).
Comparative effectiveness of the 3 intervention groups as assessed by patient satisfaction score at month 3 (End of study) | 3 months
  Patient satisfaction score will be rated using the following scale; 0=not satisfied, 1=slightly satisfied, 2= satisfied, 3=very satisfied, 4=extremely satisfied as well as patients' satisfaction questionnaire
Comparative effectiveness of the 3 intervention groups as assessed by physician global assessment at month 3 (End of study) | 3 months
  Patients will be assessed before and after treatment by one unblinded and one blinded investigators to measure the clinical improvement on a 4-point scale by comparing the photographs. The criteria for evaluation using a quartile grading scale will be as follows; 0=no improvement, 1=mild improvement (<25%), 2=moderate improvement (26% - 50%), 3=good improvement (51% -75%), 4=excellent improvement (>76%).

SECONDARY OUTCOMES:
Comparative effectiveness of the 3 intervention groups as assessed by physician global assessment at month 1 | 1 month
  Patients will be assessed before and after treatment by one unblinded and one blinded investigators to measure the clinical improvement on a 4-point scale by comparing the photographs. The criteria for evaluation using a quartile grading scale will be as follows; 0=no improvement, 1=mild improvement (<25%), 2=moderate improvement (26% - 50%), 3=good improvement (51% -75%), 4=excellent improvement (>76%).
Comparative effectiveness of the 3 intervention groups as assessed by patient global assessment at month 1 | 1 month
  Patients will be assessed before and after treatment by one unblinded and one blinded investigators to measure the clinical improvement on a 4-point scale by comparing the photographs. The criteria for evaluation using a quartile grading scale will be as follows; 0=no improvement, 1=mild improvement (<25%), 2=moderate improvement (26% - 50%), 3=good improvement (51% -75%), 4=excellent improvement (>76%).
Comparative effectiveness of the 3 intervention groups as assessed by patient satisfaction score at month 1 | 1 month
  Patient satisfaction score will be rated using the following scale; 0=not satisfied, 1=slightly satisfied, 2= satisfied, 3=very satisfied, 4=extremely satisfied as well as patients' satisfaction questionnaire
Comparative tolerability of the 3 intervention groups as assessed by the incidence of side effects (edema, pain, erythema, itching, peeling) | 3 months
  Percentage of incidence of side effects (edema, pain, erythema, itching, start of peeling) in all patients
Comparative tolerability of the fractional CO2 versus combined fractional and LLLT as regards duration of side effects in days after each laser session (edema, pain, erythema, itching, peeling) | 3 months
  Comparative tolerability of the fractional CO2 versus combined fractional and LLLT as regards duration of side effects in days after each laser session (edema, pain, erythema, itching, peeling)

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Mahgoub, MD, Principal Investigator — Cairo University; Vanessa Hafez, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr El Ainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication, as well as protocol and statistical plan analysis, are to be published starting 6 months after the publication of summary data.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 moths after publication of summary data
Access Criteria: Data will be available for 6 months and allowed access only after approval of access requests by the principal investigators.

REFERENCES:
- [Background] Yang YJ, Lee GY. Treatment of Striae Distensae with Nonablative Fractional Laser versus Ablative CO(2) Fractional Laser: A Randomized Controlled Trial. Ann Dermatol. 2011 Nov;23(4):481-9. doi: 10.5021/ad.2011.23.4.481. Epub 2011 Nov 3. PMID 22148016
- [Background] Weiss RA, McDaniel DH, Geronemus RG, Weiss MA, Beasley KL, Munavalli GM, Bellew SG. Clinical experience with light-emitting diode (LED) photomodulation. Dermatol Surg. 2005 Sep;31(9 Pt 2):1199-205. doi: 10.1111/j.1524-4725.2005.31926. PMID 16176771
- [Background] Hamblin MR. Mechanisms and applications of the anti-inflammatory effects of photobiomodulation. AIMS Biophys. 2017;4(3):337-361. doi: 10.3934/biophy.2017.3.337. Epub 2017 May 19. PMID 28748217
- [Background] Farivar S, Malekshahabi T, Shiari R. Biological effects of low level laser therapy. J Lasers Med Sci. 2014 Spring;5(2):58-62. PMID 25653800
- [Background] Cho S, Park ES, Lee DH, Li K, Chung JH. Clinical features and risk factors for striae distensae in Korean adolescents. J Eur Acad Dermatol Venereol. 2006 Oct;20(9):1108-13. doi: 10.1111/j.1468-3083.2006.01747.x. PMID 16987267
- [Background] K. Sawhney, Mossum & Hamblin, Michael. (2014). Low-level light therapy (LLLT) for cosmetics and dermatology. Progress in Biomedical Optics and Imaging - Proceedings of SPIE. 8932. 10.1117/12.2041330.
- [Background] Aldahan AS, Shah VV, Mlacker S, Samarkandy S, Alsaidan M, Nouri K. Laser and Light Treatments for Striae Distensae: A Comprehensive Review of the Literature. Am J Clin Dermatol. 2016 Jun;17(3):239-56. doi: 10.1007/s40257-016-0182-8. PMID 26923916
- [Background] Ross NA, Ho D, Fisher J, Mamalis A, Heilman E, Saedi N, Jagdeo J. Striae Distensae: Preventative and Therapeutic Modalities to Improve Aesthetic Appearance. Dermatol Surg. 2017 May;43(5):635-648. doi: 10.1097/DSS.0000000000001079. PMID 28375972
- [Background] Mishra V, Miller L, Alsaad SM, Ross EV. The Use of a Fractional Ablative Micro-Plasma Radiofrequency Device in Treatment of Striae. J Drugs Dermatol. 2015 Nov;14(11):1205-8. PMID 26580868
- [Background] Ibrahim ZA, El-Tatawy RA, El-Samongy MA, Ali DA. Comparison between the efficacy and safety of platelet-rich plasma vs. microdermabrasion in the treatment of striae distensae: clinical and histopathological study. J Cosmet Dermatol. 2015 Dec;14(4):336-46. doi: 10.1111/jocd.12160. Epub 2015 Jul 6. PMID 26147455
- [Background] Mazzarello V, Farace F, Ena P, Fenu G, Mulas P, Piu L, Rubino C. A superficial texture analysis of 70% glycolic acid topical therapy and striae distensae. Plast Reconstr Surg. 2012 Mar;129(3):589e-590e. doi: 10.1097/PRS.0b013e3182419c40. No abstract available. PMID 22374035
- [Background] Ud-Din S, McAnelly SL, Bowring A, Whiteside S, Morris J, Chaudhry I, Bayat A. A double-blind controlled clinical trial assessing the effect of topical gels on striae distensae (stretch marks): a non-invasive imaging, morphological and immunohistochemical study. Arch Dermatol Res. 2013 Sep;305(7):603-17. doi: 10.1007/s00403-013-1336-7. Epub 2013 Apr 12. PMID 23579949
- [Background] Elson, M. (1994). Topical tretinoin in the treatment of striae distensae and in the promotion of wound healing: A review. Journal of Dermatological Treatment, 5(3), 163-165. doi:10.3109/09546639409084563
- [Background] Watson RE, Parry EJ, Humphries JD, Jones CJ, Polson DW, Kielty CM, Griffiths CE. Fibrillin microfibrils are reduced in skin exhibiting striae distensae. Br J Dermatol. 1998 Jun;138(6):931-7. doi: 10.1046/j.1365-2133.1998.02257.x. PMID 9747352
- [Background] Lee KS, Rho YJ, Jang SI, Suh MH, Song JY. Decreased expression of collagen and fibronectin genes in striae distensae tissue. Clin Exp Dermatol. 1994 Jul;19(4):285-8. doi: 10.1111/j.1365-2230.1994.tb01196.x. PMID 7955466
- [Background] Sheu HM, Yu HS, Chang CH. Mast cell degranulation and elastolysis in the early stage of striae distensae. J Cutan Pathol. 1991 Dec;18(6):410-6. doi: 10.1111/j.1600-0560.1991.tb01376.x. PMID 1774350
- [Background] Gilmore SJ, Vaughan BL Jr, Madzvamuse A, Maini PK. A mechanochemical model of striae distensae. Math Biosci. 2012 Dec;240(2):141-7. doi: 10.1016/j.mbs.2012.06.007. Epub 2012 Jul 14. PMID 22796062
- [Background] Hague A, Bayat A. Therapeutic targets in the management of striae distensae: A systematic review. J Am Acad Dermatol. 2017 Sep;77(3):559-568.e18. doi: 10.1016/j.jaad.2017.02.048. Epub 2017 May 24. PMID 28551068
- [Derived] Hafez V, Mahgoub D, Satour EMA, Mikhail MMS, El-Kalioby M. Photobiomodulation versus fractional carbon dioxide laser for stria alba in phototype III-IV: a randomized controlled study. Lasers Med Sci. 2024 Jun 19;39(1):159. doi: 10.1007/s10103-024-04107-x. PMID 38890186
- See also: Low level light therapy device — http://www.fimadelettromedicali.it/site/index.php?option=com_content&view=article&id=80:laser-hpl-16-e-hpl-32-laser-ad-alta-potenza&catid=62:elettrocardiografi-ecg&Itemid=81